CLINICAL TRIAL: NCT01852747
Title: Actifuse ABX and Local Bone Have Comparable Outcomes to Local Bone in Instrumented Multi-Level Adult Spinal Deformity Patients
Brief Title: Comparison of Actifuse ABX and Local Bone in Spinal Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The sponsor merged with another company and decided they did not want to continue with the study.
Sponsor: Ohio State University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Safdar Khan, Safdar Khan, MD, Ohio State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013H0023
Record Dates: First submitted 2013-04-30; First posted 2013-05-14 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2014-02

CONDITIONS: Scoliosis; Kyphosis; Lordosis
Keywords: Spinal Deformity; Multilevel; Posterior; Lumbar; Fusion; Levoscoliosis; Dextroscoliosis; Graft
MeSH Terms: conditions — Scoliosis; Kyphosis; Lordosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multilevel Spinal Fusion w/ Actifuse ABX® (Experimental): An osteostimulatory,phase pure,porous,silicate substituted calcium phosphate bone graft substitute used during multilevel spinal fusion.
  Interventions: Procedure: Multilevel Spinal fusion with Actifuse ABX®
- Multilevel Spinal Fusion (No Intervention): Multilevel spinal fusion without Actifuse ABX.

INTERVENTIONS:
Procedure: Multilevel Spinal fusion with Actifuse ABX® — Multilevel spinal fusion as treatment for adult spinal deformity with Actifuse ABX®. Actifuse ABX® is a silicate substituted calcium phosphate bone void filler intended for orthopedic applications such as a filler for gaps and voids that are not intrinsic to the stability of the bony structure.
  Arms: Multilevel Spinal Fusion w/ Actifuse ABX®

SUMMARY:
This study is being done to compare people who had a standard of care spinal fusion using part of their local bone graft (a small amount of bone from the region of the spine where the fusion is occurring) to correct an adult spinal deformity and people who will have a standard of care spinal fusion using a mixture of Actifuse ABX® (a market approved bone graft substitute) and a local bone graft (a small amount of bone from the region of the spine where the fusion is occurring). This study will compare the outcomes of both groups to help the Orthopaedic surgeon conducting spinal fusions in the future. Investigators expect that Actifuse ABX® will be as good if not better than just a local bone graft.

DETAILED DESCRIPTION:
The current method for posterolateral lumbar fusion surgeries utilizes autograft bone typically derived from the patient's iliac crest. However, complications have been reported concerning the use of iliac crest bone, that include additional healing time due to the secondary surgical site and gait abnormalities. Clinicians are in need of an adequate alternative, and many have begun testing growth factors or synthetic compounds used in conjunction with local bone autografts. Though this avoids the need for a secondary surgical site, synthetic materials are not without their own limitations. These compounds must achieve similar growth and fusion rates as native bone. This study will test the applicability of Actifuse, a synthetic bone graft substitute, in instrumented multi-level adult spinal deformity surgery.

Actifuse is a silicate substituted calcium phosphate. It is osteostimulative, and is a bone void filler intended for orthopedic applications such as a filler for gaps and voids that are not intrinsic to the stability of the bony structure. Actifuse has several features that mimic human bone (amount of silicon, resorption rate, etc). It provides a scaffold for long-term bone healing and is intended to be packed gently into bony voids or gaps of the skeletal system, i.e. extremities, pelvis and spine including use in posterolateral spinal fusion procedures with appropriate stabilizing hardware. These defects may be surgically created osseous defects or osseous defects created from traumatic injury to the bone. The product provides a bone void filler that is resorbed and replaced by native bone during the healing process.

Actifuse accelerates bone growth by combining an interconnected macro- and micro- porous structure with osteostimulative chemistry created through a patented silicate substitution process to attach and stimulate osteoprogenitor cells (OPCs) and mesenchymal stem cells (MSCs). It resists irrigation and can be easily viewed on x-rays to monitor healing. Previous groups have shown that Actifuse is successful in the laboratory as well as in patients; however, previously reported literature has not studied the efficacy of Actifuse in instrumented multi-level adult spinal deformity.

Based on previous literature, investigators expect the Actifuse ABX to successfully fuse to native bone growth and promote fusion as well as an autograft replacement. Potential pitfalls include Actifuse not functioning as well in place of native bone. If this occurs, investigators will conduct revision surgery to ensure proper bone union.

The success of this project could have significant effects for the society at large. It is estimate that over 200,000 arthrodeses are performed each year, and the autologous iliac crest bone graft is often considered the standard of care, therefore these results could improve the outcome of surgery for thousands of patients every year. In addition, it will likely cut down on time the surgeon is in the operating room. It could also speed patient recovery by 1) lowering the amount of autologous bone harvested from the patient, and 2) taking advantage of the properties of Actifuse (osteostimulation, resorption rate, etc) that should result in quicker bone fusing and healing.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 80
* Patient received primary diagnosis of adult spinal deformity (with fusion of >2 levels)
* Patient is a candidate for multi-level posterior lumbar fusion
* Patients that do not meet any of the exclusion criteria

Exclusion Criteria:

* Non-English speaker
* Current Smoker
* Prisoner
* Patient with any of the following:

Severe degenerative disease Inflammatory bone disease (e.g. osteomyelitis) Metabolic bone disease Radiation bone therapy Existing acute or chronic infections Abnormal calcium metabolism Hypocalcaemia Severe vascular or neurological disease Cardiovascular disease precluding elective surgery Uncontrolled diabetes Severely impaired renal function Documented renal disease Malignant tumors Pregnant or nursing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Decrease patient recovery time | 12 months
  The investigators anticipate the Actifuse ABX® will decrease patient recovery time by 1) lowering the amount of autologous bone harvested from the patient and 2) taking advantage of the properties of Actifuse (osteostimulation, resorption rate, etc) that should result in quicker bone fusing and healing.

CONTACTS AND LOCATIONS:
Overall Officials: Safdar Khan, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States